CLINICAL TRIAL: NCT01797211
Title: Mediterranean Diet and Endothelial Function in Obese and Overweight Patients: the Role of Olive Oil, Non Fried Fish and Nuts
Brief Title: Mediterranean Diet and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, prof. Marco Matteo Ciccone, Associate Professor, University of Bari
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Cardiovascular Diseases
Keywords: Mediterranean diet; FMD; obesity; cardiovascular risk.
MeSH Terms: conditions — Cardiovascular Diseases; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- diet group A (Experimental): Mediterranean diet+olive oil
  Interventions: Dietary Supplement: Mediterranean diet
- Diet Group B (Experimental): Mediterranean diet+not-fried fish
  Interventions: Dietary Supplement: Mediterranean diet
- Diet Group C (Experimental): Mediterranean diet+nuts
  Interventions: Dietary Supplement: Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — Patients underwent administration of Mediterranean diet and olive oil, or Mediterranean diet and not-fried fish, or Mediterranean diet and nuts.

SUMMARY:
To assess the effect of Mediterranean diet and some of its specific components (olive oil, non fried fish and nuts) on endothelial function in overweight and obese patients

DETAILED DESCRIPTION:
Abdominal obesity is well known to increase the risk of cardiovascular disease (CVD), since it is commonly associated with hypertension, dyslipidemia, impaired fasting glucose, type 2 diabetes, metabolic syndrome, insulin resistance, systemic inflammation and endothelium dysfunction.

Abnormal endothelial function, expressed as lower vasodilatation through flow-mediated vasodilatation (FMD) of brachial artery in response to an increase in blood flow, is considered an index of subclinical atherosclerosis, and an early hallmark of cardiovascular disease, with a strong prognostic value for future cardiovascular events. Changes in diet, level of physical activity and behavior are well known key elements influence endothelial function. Recent studies seem to show that Mediterranean diet has beneficial role on cardiovascular risk. It could protect against the development of coronary heart disease also through a possible effect on body weight and obesity.

At the best of our knowledge, the effect of Mediterranean diet on endothelial function in obese subjects has not been definitely established. Therefore, the aim of this study was to evaluate the impact of Mediterranean diet on anthropometric parameters (body weight, BMI and waist circumference), lipid profile [total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C)], triglycerides (TG), fasting glucose and endothelium function, evaluated by FMD, in a group of obese and overweight subjects. In particular, subjects were invited to follow a standard Mediterranean diet for a short (3 months) or a longer (18 months) period. The specific role of some components of Mediterranean diet (olive oil or non fried fish or nuts) was also investigated.

ELIGIBILITY:
Inclusion Criteria:

BMI: > 25.0 kg/m2 Age between 18-70 years

Exclusion Criteria:

BMI < 25.0 kg/m2 Age <18 or >70 years low left ventricular ejection fraction (LVEF < 50%) symptomatic cardiac disease in advanced stage or poorly controlled by medication cerebral disorders major liver and kidney diseases cancer excessive alcohol intake use of drugs addressed to lose weight.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
3 months outcome (composite outcome) | 3 months after enrollment
  Anthropometric parameters (BMI, waist circumference [WC] and weight) a significant decrease, while FMD ones showed a significant increase after 3 months of Mediterranean diet as compared to baseline levels. The addition per se of olive oil or non fried fish or nuts to the standard Mediterranean diet did not influence anthropometric parameters, since BMI, WC and body weight of groups A, B and C were not significant different from those of the control group. After 3 months, FMD was not higher wether olive oil or non fried fish or nuts were added to standard Mediterranean diet.

SECONDARY OUTCOMES:
18 months follow-up evaluations (composite outcome) | 18 months after enrollment period
  After 18 months of dietary treatment, we observed a significant increase of HDL-C, a decrease of TC and LDL-C, no differences in TG plasma concentrations and fasting glucose. The addition per se of olive oil or non fried fish or nuts to the standard Mediterranean diet did not influence the lipid profile. Anthropometric parameters showed a significant decrease and FMD showed a significant increase after 18 months, as compared to 3 months levels. Olive oil, non fried fish or nuts to the standard Mediterranean diet did not influence anthropometric parameters, since BMI, WC and body weight of groups A, B and C were not significant different from those of the control group. It is noteworthy that, after 18 months of Mediterranean diet, but not after 3 months, FMD was higher wether olive oil or non fried fish or nuts were added to standard Mediterranean diet. Lastly, at 18 months, the FMD levels of groups A, B, and C were significantly higher than those of control group.

CONTACTS AND LOCATIONS:
Overall Officials: Marco M Ciccone, MD, Principal Investigator — University of Bari; Giovanni De Pergola, MD, Principal Investigator — University of Bari
Locations (1):
- Section of Cardiovascular Diseases, Department of Emergency and Organ Transplantation, University of Bari, Bari, Bari, Italy

REFERENCES:
- [Background] Feletou M, Vanhoutte PM. Endothelium-derived hyperpolarizing factor: where are we now? Arterioscler Thromb Vasc Biol. 2006 Jun;26(6):1215-25. doi: 10.1161/01.ATV.0000217611.81085.c5. Epub 2006 Mar 16. PMID 16543495
- [Background] Yoshida T, Kawano H, Miyamoto S, Motoyama T, Fukushima H, Hirai N, Ogawa H. Prognostic value of flow-mediated dilation of the brachial artery in patients with cardiovascular disease. Intern Med. 2006;45(9):575-9. doi: 10.2169/internalmedicine.45.1534. Epub 2006 Jun 1. PMID 16755087
- [Result] Kastorini CM, Milionis HJ, Goudevenos JA, Panagiotakos DB. Mediterranean diet and coronary heart disease: is obesity a link? - A systematic review. Nutr Metab Cardiovasc Dis. 2010 Sep;20(7):536-51. doi: 10.1016/j.numecd.2010.04.006. PMID 20708148
- [Result] Babio N, Bullo M, Basora J, Martinez-Gonzalez MA, Fernandez-Ballart J, Marquez-Sandoval F, Molina C, Salas-Salvado J; Nureta-PREDIMED Investigators. Adherence to the Mediterranean diet and risk of metabolic syndrome and its components. Nutr Metab Cardiovasc Dis. 2009 Oct;19(8):563-70. doi: 10.1016/j.numecd.2008.10.007. Epub 2009 Jan 26. PMID 19176282
- [Result] Jambrik Z, Venneri L, Varga A, Rigo F, Borges A, Picano E. Peripheral vascular endothelial function testing for the diagnosis of coronary artery disease. Am Heart J. 2004 Oct;148(4):684-9. doi: 10.1016/j.ahj.2004.04.016. PMID 15459601
- [Result] Wildman RP, Muntner P, Reynolds K, McGinn AP, Rajpathak S, Wylie-Rosett J, Sowers MR. The obese without cardiometabolic risk factor clustering and the normal weight with cardiometabolic risk factor clustering: prevalence and correlates of 2 phenotypes among the US population (NHANES 1999-2004). Arch Intern Med. 2008 Aug 11;168(15):1617-24. doi: 10.1001/archinte.168.15.1617. PMID 18695075
- [Result] Hotchkiss JW, Leyland AH. The relationship between body size and mortality in the linked Scottish Health Surveys: cross-sectional surveys with follow-up. Int J Obes (Lond). 2011 Jun;35(6):838-51. doi: 10.1038/ijo.2010.207. Epub 2010 Oct 5. PMID 20921963
- [Result] von Ruesten A, Steffen A, Floegel A, van der A DL, Masala G, Tjonneland A, Halkjaer J, Palli D, Wareham NJ, Loos RJ, Sorensen TI, Boeing H. Trend in obesity prevalence in European adult cohort populations during follow-up since 1996 and their predictions to 2015. PLoS One. 2011;6(11):e27455. doi: 10.1371/journal.pone.0027455. Epub 2011 Nov 10. PMID 22102897
- [Result] Serdula MK, Mokdad AH, Williamson DF, Galuska DA, Mendlein JM, Heath GW. Prevalence of attempting weight loss and strategies for controlling weight. JAMA. 1999 Oct 13;282(14):1353-8. doi: 10.1001/jama.282.14.1353. PMID 10527182
- [Result] Romaguera D, Norat T, Vergnaud AC, Mouw T, May AM, Agudo A, Buckland G, Slimani N, Rinaldi S, Couto E, Clavel-Chapelon F, Boutron-Ruault MC, Cottet V, Rohrmann S, Teucher B, Bergmann M, Boeing H, Tjonneland A, Halkjaer J, Jakobsen MU, Dahm CC, Travier N, Rodriguez L, Sanchez MJ, Amiano P, Barricarte A, Huerta JM, Luan J, Wareham N, Key TJ, Spencer EA, Orfanos P, Naska A, Trichopoulou A, Palli D, Agnoli C, Mattiello A, Tumino R, Vineis P, Bueno-de-Mesquita HB, Buchner FL, Manjer J, Wirfalt E, Johansson I, Hellstrom V, Lund E, Braaten T, Engeset D, Odysseos A, Riboli E, Peeters PH. Mediterranean dietary patterns and prospective weight change in participants of the EPIC-PANACEA project. Am J Clin Nutr. 2010 Oct;92(4):912-21. doi: 10.3945/ajcn.2010.29482. Epub 2010 Sep 1. PMID 20810975
- [Result] Issa C, Darmon N, Salameh P, Maillot M, Batal M, Lairon D. A Mediterranean diet pattern with low consumption of liquid sweets and refined cereals is negatively associated with adiposity in adults from rural Lebanon. Int J Obes (Lond). 2011 Feb;35(2):251-8. doi: 10.1038/ijo.2010.130. Epub 2010 Jul 6. PMID 20603626
- [Result] de Lorgeril M, Salen P, Martin JL, Monjaud I, Delaye J, Mamelle N. Mediterranean diet, traditional risk factors, and the rate of cardiovascular complications after myocardial infarction: final report of the Lyon Diet Heart Study. Circulation. 1999 Feb 16;99(6):779-85. doi: 10.1161/01.cir.99.6.779. PMID 9989963
- [Result] Robertson RM, Smaha L. Can a Mediterranean-style diet reduce heart disease? Circulation. 2001 Apr 3;103(13):1821-2. doi: 10.1161/01.cir.103.13.1821. No abstract available. PMID 11282917
- [Result] Perona JS, Cabello-Moruno R, Ruiz-Gutierrez V. The role of virgin olive oil components in the modulation of endothelial function. J Nutr Biochem. 2006 Jul;17(7):429-45. doi: 10.1016/j.jnutbio.2005.11.007. Epub 2005 Dec 12. PMID 16481154
- [Result] Massaro M, Basta G, Lazzerini G, Carluccio MA, Bosetti F, Solaini G, Visioli F, Paolicchi A, De Caterina R. Quenching of intracellular ROS generation as a mechanism for oleate-induced reduction of endothelial activation and early atherogenesis. Thromb Haemost. 2002 Aug;88(2):335-44. PMID 12195709
- [Result] Tuck KL, Hayball PJ. Major phenolic compounds in olive oil: metabolism and health effects. J Nutr Biochem. 2002 Nov;13(11):636-644. doi: 10.1016/s0955-2863(02)00229-2. PMID 12550060
- [Result] Levitan EB, Wolk A, Mittleman MA. Fish consumption, marine omega-3 fatty acids, and incidence of heart failure: a population-based prospective study of middle-aged and elderly men. Eur Heart J. 2009 Jun;30(12):1495-500. doi: 10.1093/eurheartj/ehp111. Epub 2009 Apr 21. PMID 19383731
- [Result] Shah AP, Ichiuji AM, Han JK, Traina M, El-Bialy A, Meymandi SK, Wachsner RY. Cardiovascular and endothelial effects of fish oil supplementation in healthy volunteers. J Cardiovasc Pharmacol Ther. 2007 Sep;12(3):213-9. doi: 10.1177/1074248407304749. PMID 17875948
- [Result] Anderson JS, Nettleton JA, Herrington DM, Johnson WC, Tsai MY, Siscovick D. Relation of omega-3 fatty acid and dietary fish intake with brachial artery flow-mediated vasodilation in the Multi-Ethnic Study of Atherosclerosis. Am J Clin Nutr. 2010 Nov;92(5):1204-13. doi: 10.3945/ajcn.2010.29494. Epub 2010 Sep 8. PMID 20826628
- [Result] Kelly JH Jr, Sabate J. Nuts and coronary heart disease: an epidemiological perspective. Br J Nutr. 2006 Nov;96 Suppl 2:S61-7. doi: 10.1017/bjn20061865. PMID 17125535
- [Result] Sabate J, Ang Y. Nuts and health outcomes: new epidemiologic evidence. Am J Clin Nutr. 2009 May;89(5):1643S-1648S. doi: 10.3945/ajcn.2009.26736Q. Epub 2009 Mar 25. PMID 19321572
- [Result] Urpi-Sarda M, Casas R, Chiva-Blanch G, Romero-Mamani ES, Valderas-Martinez P, Arranz S, Andres-Lacueva C, Llorach R, Medina-Remon A, Lamuela-Raventos RM, Estruch R. Virgin olive oil and nuts as key foods of the Mediterranean diet effects on inflammatory biomakers related to atherosclerosis. Pharmacol Res. 2012 Jun;65(6):577-83. doi: 10.1016/j.phrs.2012.03.006. Epub 2012 Mar 18. PMID 22449789
- [Result] Hamdy O. Lifestyle modification and endothelial function in obese subjects. Expert Rev Cardiovasc Ther. 2005 Mar;3(2):231-41. doi: 10.1586/14779072.3.2.231. PMID 15853597